CLINICAL TRIAL: NCT02442089
Title: Health Call: A Randomized Control Trial of Interactive Automated Reminder Calls to Reduce Failure to Attend Rates at an Urban Referral Hospital in Chile
Brief Title: Impact of Automated Calls on Pediatric Patient Attendance in Chile
Acronym: Health Call
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Hospital Luis Calvo Mackenna (Unknown); Merlin Telecom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00004109
Record Dates: First submitted 2015-04-06; First posted 2015-05-13 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2015-05

CONDITIONS: Attendance
Keywords: mHealth; eHealth; Health Systems; Health Technology; No Show; Non-attendance; Chile; Randomized controlled trial; Efficiency, Organizational; Pediatric Hospitals; Global Health; Referral and Consultation; Health Care Systems; Community Health Systems; Health Information Systems; Integrated Health Care Systems; Community Medicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention (No Intervention): The intervention arm subjects will not receive the automated interactive voice reminder before their appointment.
- Intervention (Experimental): The intervention arm subjects will receive the automated interactive voice reminder before their appointment.
  Interventions: Behavioral: Health Call

INTERVENTIONS:
Behavioral: Health Call — Health Call is an automated interactive voice reminder system that can contact guardians of patients ahead of their child's appointment, asks then confirms a security question about the patient, then, if the call recipient passes the security screen, provides a reminder about upcoming appointment.
  Arms: Intervention

SUMMARY:
Missed health care appointments present a serious challenge to patient care. Especially in government funded health systems like that of Chile, missed appointments can lead to delayed care, wasted resources, and escalating costs.

This private-public-research collaboration seeks to provide a rigorous, practical evaluation of a new patient reminder system, evaluate how health beliefs impact patient attendance, and capture the potential for scaling up this or other health technology systems. Using a mixed-methods approach this study will provide contextualized, triangulated analysis of pediatric patient attendance in Chile.

DETAILED DESCRIPTION:
The Health Call study is divided into two phases. The first phase is a randomized controlled trial and side-by- side cost-benefit analysis. Enrolled guardians of pediatric patients will complete a questionnaire at the point of referral and then be randomized to intervention, the automated reminder system, or no reminder. The investigators will then monitor attendance status at their subsequent appointment and evaluate whether the appointment reminders affected attendance as well as the cost-benefit ratio of using the reminder system.

The second phase will involve interviewing guardians and healthcare professionals. These interviews have two foci. First, combined with patient, guardian, and/or household data from the randomized trial, these results will be used to develop a more comprehensive understanding of why pediatric patients attend appointments. The second focus is on improving the reminder system and developing new health technology interventions that can increase patient attendance.

ELIGIBILITY:
Inclusion Criteria:

* Guardian with a phone number (land-line or mobile) who is able to receive and answer voice calls
* Guardian who is willing to take part in the study and complete the consent form
* Guardian who is sufficiently proficient in Spanish so as to complete the questionnaire
* Guardian's patient who has a referral appointment at Hospital Luis Calvo Mackenna who is 18 years of age or younger

Exclusion Criteria:

* Guardian or child who do not meet the inclusion criteria
* Anyone that lives in the same household as an enrolled study participant.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 263 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Intervention impact | 9 months
  Evaluate whether a patient reminder system, Health Call, can decrease the overall failure to attend appointment rate as a percentage of overall appointments
Key attendance factors | 9 months
  Examine what demographic or health belief factors are significantly related to appointment attendance as measured by a psychometric questionnaire
Develop new interventions | 9 months
  Investigate staff and recipient opinions of patient attendance, the Health Call system, and ideas for future interventions to reduce failure to attend as measured through in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: William Weiss, DrPH, MA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Hospital Luis Calvo Mackenna, Santiago, Chile